CLINICAL TRIAL: NCT07345676
Title: Optimizing Evidence-Based Interventions to Improve Colorectal Cancer Screening Adherence in Community Health Clinics
Brief Title: Colorectal Cancer Screening Outreach
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Yale University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Screening
Other Study IDs: 2000041322
Record Dates: First submitted 2026-01-07; First posted 2026-01-16 (Actual); Last update posted 2026-02-09 (Actual); Status verified 2026-02

CONDITIONS: Colo-rectal Cancer
Keywords: Screening adherence
MeSH Terms: conditions — Colonic Neoplasms

STUDY DESIGN:
Intervention Model Description: The study will include adults who receive care at a local, multisite federally qualified health center, who have outstanding orders for colorectal cancer screening.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Control-Usual Care (No Intervention): Participants will receive a simple text message reminder
- Messaging Group A (Experimental): Participants will receive a series of outreach messages including texts with two-way messaging capabilities, mailed letter, and a reminder to their clinician. Content of the text message arm will be varied so that patients receive one of three messages (A, B or C).
  Interventions: Behavioral: Bundled messaging intervention
- Messaging Group B (Experimental): Participants will receive a series of outreach messages including texts with two-way messaging capabilities, mailed letter, and a reminder to their clinician. Content of the text message arm will be varied so that patients receive one of three messages (A, B or C).
  Interventions: Behavioral: Bundled messaging intervention
- Messaging Group C (Experimental): Participants will receive a series of outreach messages including texts with two-way messaging capabilities, mailed letter, and a reminder to their clinician. Content of the text message arm will be varied so that patients receive one of three messages (A, B or C).
  Interventions: Behavioral: Bundled messaging intervention

INTERVENTIONS:
Behavioral: Bundled messaging intervention — A bundled intervention of text message, letter, and provider reminder. Text message content using behaviorally motivated messages will vary.
  Arms: Messaging Group A; Messaging Group B; Messaging Group C

SUMMARY:
This is a 4 arm pragmatic trial to test a multicomponent intervention designed to improve adherence to colorectal cancer screening.

ELIGIBILITY:
Inclusion Criteria:

* Established adult medicine patient at Cornell Scott Hill health (defined as having a CSHH primary care doctor or >1 adult medicine visits in the last year).
* Incomplete colorectal cancer screening test defined as an outstanding order for colonoscopy or stool-based CRC screening (e.g., fecal immunochemical test (FIT) or FIT-DNA testing), but no evidence of test completion at the time of randomization. Orders must have been placed between 90-180 days prior to randomization.

OR

* Abnormal stool-based test without follow-up, defined as an abnormal stool-based test result (e.g., positive FIT or FIT-DNA) with no completed diagnostic colonoscopy within 90 days of the result. Patients who meet this criterion will be included in a non randomized arm of the study.

Exclusion Criteria:

* Because this is a pragmatic study of a behavioral intervention to improve colorectal cancer screening adherence, any participants who otherwise meet the inclusion criteria will not be excluded.

Ages: 45 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2000 (Estimated)
Dates: Start 2026-03 (Estimated); Primary Completion 2027-01 (Estimated); Study Completion 2027-04 (Estimated)

PRIMARY OUTCOMES:
Number of participants with scheduled or completed colorectal cancer screening. | up to 3 months from randomization
  Number of participants who completed or scheduled screening (colonoscopy or stool-based test) within 3 months of randomization.

SECONDARY OUTCOMES:
Number of participants with abnormal stool-based test that complete a diagnostic colonoscopy. | up to 90 days from intervention
  Number of participants with abnormal stool-based test who complete a diagnostic colonoscopy within 90 days of intervention.
Number of participants who complete screening. | up to 90 days from randomization
  Number of participants who complete screening (stool-based testing or colonoscopy) within 90 days of randomization.
Number of participants who achieve the primary endpoint. | 6 months post randomization
  Number of participants who achieve the primary endpoint (screening or scheduling of screening) at 6 months post randomization.
Number of participants who achieve the primary endpoint by message type. | up to 90 days from randomization
  Number of participants who achieve the primary endpoint (screening scheduling or completion rate at 90 days) by message type (message A/B/C).
Number of participants who complete screening within 6 months of initial outreach. | up to 6 months from initial outreach
  Number of participants who complete screening within 6 months of initial outreach by text message type (message A/B/C).
Number of participants who complete screening colonoscopy within 6 months of initial outreach. | up to 6 months from initial outreach
  Number of participants who complete screening colonoscopy within 6 months of initial outreach by text message type (message A/B/C).
Number of participants who provide any response. | 7, 14, 21, and 90 days
  Number of participants who provide any response to text messages by message type (message A/B/C).
Number of participants who achieve the primary outcome from among those who did and did not respond to any text message. | 6 months post randomization
  Number of participants who achieve the primary outcome from among those who did and did not respond to any text message.
Number of providers who respond to reminders. | 6 months post randomization
  Number of providers who respond to provider reminders through MyChart message, phone call, or in-clinic discussion.

CONTACTS AND LOCATIONS:
Overall Officials: Ilana Richman, MD, Principal Investigator — Yale University
Locations (1):
- Cornell Scott Hill Health, New Haven, Connecticut, United States

IPD SHARING:
Plan to Share IPD: No